CLINICAL TRIAL: NCT03579472
Title: A Phase Ib Trial of M7824 and Eribulin in Patients With Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: M7824 and Eribulin Mesylate in Treating Patients With Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the fact that the sponsor decided not to move forward with the development of M7824
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0500; NCI-2018-01140 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0500 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-07-06 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — bintrafusp alfa protein, human; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bintrafusp alfa, eribulin mesylate) (Experimental): Patients receive bintrafusp alfa IV over 50-80 minutes on days 1, 15, and 29, and eribulin mesylate IV over 2-5 minutes on days 1, 8, 22, and 29. Treatment repeats every 42 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog

SUMMARY:
This phase Ib trial studies the best dose and side effects of eribulin mesylate when given together with M7824)in treating patients with triple negative breast cancer that has spread to other places in the body. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as M7824, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving eribulin mesylate and M7824 may work better at treating triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of eribulin mesylate (eribulin) when in combination with the fixed dose of bintrafusp alfa (M7824) in patients with metastatic triple-negative breast cancer (TNBC).

II. To evaluate the safety and tolerability of M7824 when in combination with eribulin in patients with metastatic TNBC.

SECONDARY OBJECTIVES:

I. To determine the best overall response (BOR) rate according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To determine the overall response rate (ORR).

OTHER OBJECTIVES:

I. To assess immunologic/molecular responses to M7824 in combination with eribulin in patients with metastatic TNBC.

II. Estimation of progression-free survival (PFS) in metastatic TNBC patients treated with M7824 in combination with eribulin.

III. Perform correlative studies on blood and tissue samples to evaluate systemic and tumor biomarkers of response and resistance to M7824 and eribulin.

IV. Correlative studies on blood and tissue samples will also be used to evaluate systemic and tumor biomarkers of response to M7824 and eribulin.

OUTLINE:

Patients receive bintrafusp alfa intravenously (IV) over 50-80 minutes on days 1, 15, and 29, and eribulin mesylate IV over 2-5 minutes on days 1, 8, 22, and 29. Treatment repeats every 42 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Histologically confirmed metastatic triple negative breast cancer with measurable disease by RECIST 1.1 criteria

  * Hormone receptor (HR) defined as positive for the purposes of this study, if expression of estrogen receptor (ER) and/or progesterone receptor (PR) expression is greater than 10% by immunohistochemistry (IHC) and HER2 negative or non-amplified is determined by the current American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) criteria, which are as follows: HER2 testing by IHC as 0 or 1+. If HER2 is 2+, ISH (in situ hybridization) must be performed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Baseline multi-gated acquisition scan (MUGA) or echocardiogram scans with left ventricular ejection fraction (LVEF) of > 50%.
* Absolute neutrophil count (ANC) >= 1500 cells/uL.
* White blood cell (WBC) counts > 2500/uL.
* Lymphocyte count >= 300/uL.
* Platelet count >= 100,000/uL.
* Hemoglobin >= 9.0 g/dL.
* Hepatic impairment Child-Pugh < B7.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) with the following exception:

  * Patients with known Gilbert disease who have serum indirect bilirubin level =< 3 X ULN may be enrolled. Eribulin dose modification will be needed in patients with hepatic insufficiency according to the US Prescribing Information (product insert)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN with the following exception: patients with liver involvement: AST and/or ALT =< 5 x ULN.
* Alkaline phosphatase =< 2.5 x ULN with the following exception: patients with documented liver involvement or bone metastases: alkaline phosphatase =< 5 x ULN.
* Creatinine clearance >= 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation.
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy during the study and for at least 4 months after the last dose of study drugs in such a manner that the risk of pregnancy is minimized. Men on study also must be using contraception. Women of childbearing potential (WOCBP) are women who have not been postmenopausal greater than 1 year or undergone a hysterectomy or bilateral oophorectomy.
* Negative serum or urine pregnancy test for women within 72 hours of receiving the first dose of the study medication for women of childbearing potential.
* Has received no more than 5 previous lines of chemotherapy in the metastatic setting.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) for metastatic breast cancer-or- if patient has had prior immune-oncology therapies in the neoadjuvant or adjuvant setting within the past 12 months.
* Has had major surgery within 21 days before cycle 1, day 1.
* Uncontrolled inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
* Serious intercurrent infections or non-malignant medical illness that are uncontrolled or the control of which may be jeopardized by this therapy.
* Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocols.
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.
* Patients with a history of autoimmune hypothyroidism (such as atrophic thyroiditis) on a stable dose of thyroid replacement hormone may be eligible.
* Patients with uncontrolled type 1 diabetes mellitus. If on a stable insulin regimen may be eligible, after discussion with principal investigator.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations.
  * Rash must cover less than 10% of body surface area (BSA).
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%). No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids).
* Patients with human immunodeficiency virus (HIV)-1 may be eligible if they meet the following conditions:

  * CD4 cell count >= 350 cells/mm^3 obtained within 90 days prior to study start.
  * Plasma HIV-1 ribonucleic acid (RNA) below detected limit obtained by Food and Drug Administration (FDA)-approved assays for > 2 years on combination anti-retroviral therapy (cART).
  * Plasma HIV-1 RNA level of less than 40 copies/mL obtained by the Abbott m2000 assay or less than 20 copies/mL by Roche Taqman version (v)2.0 assay within 90 days prior to study start.
  * Plasma HIV-1 RNA greater than or equal to 0.4 copies/mL by single copy assay within 120 days prior to entry.
  * Receiving a stable cART regimen containing at least 3 agents (not including ritonavir if less than a 200 mg total daily dose) with no change in the components of antiretroviral therapy for at least 90 days prior to study entry.
* Patients with prior allogeneic stem cell or solid organ transplantation.
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Patients with known active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Known active tuberculosis.
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to cycle 1, day 1 or at any time during the study.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug, whichever is shorter, from cycle 1 day 1.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 1 week prior to cycle 1 day 1, or anticipated requirement for systemic immunosuppressive medications during the trial. Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone prior to the anthracycline-based chemotherapy for nausea) may be enrolled in the study. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
* Concurrent disease or condition that would interfere with study participation or safety, such as any of the following:

  * Active, clinically significant infection either grade > 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 or requiring the use of parenteral anti-microbial agents within 14 days before day 1 of study drug.
  * Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders.
  * Non-healing wound, ulcer, or bone fracture.
* Known hypersensitivity to any of the components of M7824 or eribulin.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Subjects with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention, including leptomeningeal disease, are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy.
* History of conditions associated with bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | Up to 90 days post-treatment
  Will be defined as highest dose with dose limiting toxicity (DLT) rate =< 30%. The number of patients on each dose as well as DLTs will be summarized. Bayesian optimal interval (BOIN) design will be employed to identify the RP2D of eribulin with M7824.
Incidence of adverse events | Up to 90 days post-treatment
  Safety and tolerability will be assessed in terms of adverse events (AEs), and serious adverse events (SAEs). AEs and SAEs will be tabulated using frequencies and percentages, by severity, by grade, and by relationship to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Damodaran, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org